CLINICAL TRIAL: NCT04463407
Title: Efectividad de Una intervención Educativa Preventiva Previa a Vacaciones de Fiestas Patrias Sobre la composición Corporal, hábitos de alimentación y Niveles de Actividad física en Estudiantes Universitarios: Estudio Aleatorizado Controlado
Brief Title: Effect of a Single Nutritional Intervention Previous to a Critical Period of Fat Gain in University Students With Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Valparaiso (Other)
Responsible Party: Principal Investigator, Carlos Cristi Montero, Principal Investigator, Pontificia Universidad Catolica de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIOEPUCV-H145-2017
Record Dates: First submitted 2020-06-26; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants keep their normal routine without intervention.
- Experimental group (Experimental): Participants receive a single nutritional intervention previous to a critical period.
  Interventions: Other: Educational talk about physical activity and nutritional recommendations before a critical period of fat gain in university students

INTERVENTIONS:
Other: Educational talk about physical activity and nutritional recommendations before a critical period of fat gain in university students — An intervention was performed emulating a traditional nutritional session from a primary healthcare center (public health system). Traditionally, this session lasts around 20 minutes and includes a body composition measurement, nutritional assessment, and a brief educational talk about healthy eating. Just the intervention group received a series of healthy recommendations specially focused on the National Holiday.
  Arms: Experimental group

SUMMARY:
The present study aimed to investigate the effects of a single nutritional preventive session previous to a critical period linked to fat gain in university students with overweight and obesity, emulating a nutritional session of a public health system.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [BMI] ≥25 kg/m2
* Not having metal plates
* Not studying Nutrition and Dietetics or Physical Education
* Not being pregnant

Exclusion Criteria:

- Presente gastrointestinal problems (vomit or diarrheas) during the three weeks that last the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Body composition measurements | 3 weeks
  Changes on fat mass measured by DXA

SECONDARY OUTCOMES:
Feeding questionnaires and food guide recommendations | 3 weeks
  Changes on the Global Food Index
Feeding questionnaires and food guide recommendations | 3 weeks
  Changes on the KIDMED index (questionnaire establishes the adherence to the Mediterranean diet)
Feeding questionnaires and food guide recommendations | 3 weeks
  Changes on the Food Guide Recommendation
Physical activity level | 3 weeks
  Modification on physical activity level measured by accelerometry

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education, Pontificia Universidad Católica de Valparaíso, Valparaíso, Chile, Valparaíso, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No
All participant data are private.

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT04463407/SAP_000.pdf